CLINICAL TRIAL: NCT03160859
Title: Prospective RCT of Water Exchange (WE) vs. WE Plus Cap-Assisted Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: VA Northern California Health Care System (U.S. Federal Agency); VA Palo Alto Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: GAST-015-16S; NCT03543124 (obsolete NCT alias)
Record Dates: First submitted 2017-05-12; First posted 2017-05-19 (Actual); Results first posted 2023-12-12 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-11

CONDITIONS: Unsedated Colonoscopy; Water Exchange Colonoscopy; Cap; Colonoscopy Pain
Keywords: unsedated colonoscopy; water exchange colonoscopy; cap; colonoscopy pain
MeSH Terms: conditions — Anterior polar cataract 2 | interventions — Methods

STUDY DESIGN:
Intervention Model Description: This will be a multi-VA site, prospective RCT to compare different methods with 2 arms to determine which is less painful: water alone or water plus cap. Randomization will be based on computer generated random numbers placed inside opaque sealed envelopes. The envelope will be opened to reveal the code when the colonoscopist is ready to insert the endoscope to begin the examination. Patients who are willing to participate will sign an informed consent before starting the colonoscopy procedure. Separate parallel randomization will be set up at each site. Control Method: Involves unsedated colonoscopy with water exchange. Residual air will be removed and water will be infused to guide insertion through an airless lumen. Infused water will be removed by suction, along with residual fecal debris, predominantly during insertion. Study method: Involves unsedated colonoscopy with water exchange and the addition of a commercially available accessory fitted onto the colonoscope.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Control Method (Other): One arm of the study will include unsedated colonoscopy with water exchange (WE) as the control method. Residual air in the colon will be removed and water will be infused to guide insertion through an airless lumen. Infused water will be removed predominantly during insertion.
  Interventions: Other: Control
- Study Method (Other): The other arm will include unsedated colonoscopy with water exchange (WE) and the addition of a simple commercially available accessory to the colonoscopy device: a cap (Disposable Distal Attachment, Olympus Medical Systems Corp., Tokyo, Japan) fitted to the colonoscope per manufacturer instruction. Residual air in the colon will be removed and water will be infused to guide insertion through an airless lumen. Infused water will be removed predominantly during insertion.
  Interventions: Device: Study method

INTERVENTIONS:
Other: Control — Unsedated colonoscopy with water exchange (WE) where the residual air in the colon will be removed and water will be infused to guide insertion through an airless lumen. Infused water is removed predominantly during insertion.
  Other Names: Water exchange method
  Arms: Control Method
Device: Study method — Unsedated colonoscopy with water exchange (WE + cap) and the addition of a cap fitted to the colonoscope.
  Other Names: Water exchange method plus cap
  Arms: Study Method

SUMMARY:
This is a study to compare two different, but normally, used methods of colonoscopy in patients undergoing colonoscopy without sedation. There will be two arms in this study: WE (water exchange) control, and WE (water exchange) plus cap (placed at tip of the colonoscope). The patient will prepare himself/herself for the colonoscopy as per normal instructions and he/she will be given the information for the study at that time so that he/she can make a decision to participate in the study. The control method will use water instead of air during insertion of the colonoscope. The study method will use a cap that will fit onto the end of the colonoscope plus water during insertion of the colonoscope. This study will assess if the study method is less painful than the control method.

DETAILED DESCRIPTION:
This will be a multi-VA site, unblinded investigators, prospective randomized control trial (RCT). Randomization (WE, WE + cap) will be based on computer generated random numbers placed inside opaque sealed envelopes. The envelope (in pre-arranged order set up by statistics consultant) will be opened to reveal the code when the colonoscopist is ready to insert the endoscope to begin the examination. This will be a comparison of two arms (WE, WE + cap) to see which one is less painful.

Patients who are willing to participate will sign an informed consent before starting the colonoscopy procedure. Separate parallel randomization will be set up at each site, stratified type of colonoscopy (screening, surveillance, diagnostic). All subjects will have scheduled unsedated colonoscopy as a result of lack of escort or personal preference for no sedation. Randomization will be set up by statistics consultant.

Control Method: One arm of the study will include unsedated colonoscopy with water exchange (WE) as the control method. Residual air in the colon will be removed and water will be infused to guide insertion through an airless lumen. Infused water will be removed by suction, along with residual fecal debris, predominantly during insertion.

Study method: The other arm will include unsedated colonoscopy with water exchange (WE) and the addition of a cap, fitted to the colonoscope per manufacturer instruction.

ELIGIBILITY:
Inclusion Criteria:

* Informed/educated (about pros and cons of the unsedated option) Veterans undergoing:

  * diagnostic
  * surveillance (follow up of polyps)
  * screening (first-time) colonoscopy at participating sites
  * choosing scheduled unsedated colonoscopy for any reason (lack of escort, personal preference)

Exclusion Criteria:

* decline to be randomized
* unable to give consent or respond to questionnaires
* history of colon surgery
* active inflammatory bowel disease
* lower gastrointestinal bleeding (except for occult blood or FIT positive in the context of colon cancer screening)
* therapeutic colonoscopy (e.g., hemostasis, removal of large polyp)
* proctosigmoidoscopy
* bidirectional endoscopy
* inadequate consumption of bowel preparation
* known history of severe diverticulosis or diverticulitis
* history of abdominal surgery previously requiring sedation for colonoscopy
* current narcotic/anxiolytic medication use
* prior unsuccessful experience with unsedated colonoscopy
* emergent colonoscopy
* evidence of colonic obstruction based on pre-colonoscopy clinical evaluation
* current participation in other studies
* medical condition that could increase the risk associated with colonoscopy

  * active cardiac
  * or pulmonary disease
  * or other serious disease
* medical condition that would preclude a benefit from colonoscopic screening

  * cancer
  * or any terminal illness
* prosthetic heart valve
* anticoagulant therapy
* nonmedical problems

  * psychiatric disorders
  * excessive use of alcohol
* need for special precautions in performing colonoscopy

  * antibiotic prophylaxis
* request of on demand sedation

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2018-06-08 (Actual); Primary Completion 2022-10-28 (Actual); Study Completion 2022-10-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Felix W. Leung, MD, Principal Investigator — VA Greater Los Angeles Healthcare System, Sepulveda, CA
Locations (3):
- United States (3):
  - VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California
  - VA Northern California Health Care System, Mather, CA, Sacramento, California
  - VA Greater Los Angeles Healthcare System, Sepulveda, CA, Sepulveda, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wolff WI, Shinya H. Polypectomy via the fiberoptic colonoscope. Removal of neoplasms beyond reach of the sigmoidoscope. N Engl J Med. 1973 Feb 15;288(7):329-32. doi: 10.1056/NEJM197302152880701. No abstract available. PMID 4682941
- [Background] Leung FW. The case of unsedated screening colonoscopy in the United States. Gastrointest Endosc. 2009 Jun;69(7):1354-6. doi: 10.1016/j.gie.2008.12.234. Epub 2009 Feb 27. No abstract available. PMID 19249764
- [Background] Leung FW, Aljebreen AM, Brocchi E, Chang EB, Liao WC, Mizukami T, Schapiro M, Triantafyllou K. Sedation-risk-free colonoscopy for minimizing the burden of colorectal cancer screening. World J Gastrointest Endosc. 2010 Mar 16;2(3):81-9. doi: 10.4253/wjge.v2.i3.81. PMID 21160707
- [Background] Leung FW. Is there a place for sedationless colonoscopy? J Interv Gastroenterol. 2011 Jan;1(1):19-22. doi: 10.4161/jig.1.1.14592. PMID 21686108
- [Background] Cataldo PA. Colonoscopy without sedation. Dis Colon Rectum. 1996 Mar;39(3):257-61. doi: 10.1007/BF02049463. PMID 8603544
- [Background] Hoffman MS, Butler TW, Shaver T. Colonoscopy without sedation. J Clin Gastroenterol. 1998 Jun;26(4):279-82. doi: 10.1097/00004836-199806000-00013. PMID 9649011
- [Background] Rex DK, Imperiale TF, Portish V. Patients willing to try colonoscopy without sedation: associated clinical factors and results of a randomized controlled trial. Gastrointest Endosc. 1999 May;49(5):554-9. doi: 10.1016/s0016-5107(99)70381-0. PMID 10228251
- [Background] Subramanian S, Liangpunsakul S, Rex DK. Preprocedure patient values regarding sedation for colonoscopy. J Clin Gastroenterol. 2005 Jul;39(6):516-9. doi: 10.1097/01.mcg.0000165667.79530.44. PMID 15942439
- [Background] Early DS, Saifuddin T, Johnson JC, King PD, Marshall JB. Patient attitudes toward undergoing colonoscopy without sedation. Am J Gastroenterol. 1999 Jul;94(7):1862-5. doi: 10.1111/j.1572-0241.1999.01219.x. PMID 10406249
- [Background] Leung FW. Patients' perspective - written testimonials from physician-patients and oral accounts presented by patients in person. J Interv Gastroenterol. 2011 Jan;1(1):45-46. doi: 10.4161/jig.1.1.14605. No abstract available. PMID 21686115
- [Background] Jonas DE, Russell LB, Sandler RS, Chou J, Pignone M. Patient time requirements for screening colonoscopy. Am J Gastroenterol. 2007 Nov;102(11):2401-10. doi: 10.1111/j.1572-0241.2007.01387.x. Epub 2007 Jun 29. PMID 17608779
- [Background] Leung FW. Unsedated colonoscopy introduced to ensure access is acceptable to a subgroup of veterans. Dig Dis Sci. 2008 Oct;53(10):2719-22. doi: 10.1007/s10620-007-0192-8. Epub 2008 Feb 15. PMID 18274901
- [Background] Felix W. Leung, Hartley Cohen, Stanley K. Dea, Dennis M. Jensen, Thomas O. Kovacs, Gordon V. Ohning, Joseph R. Pisegna, Alireza Sedarat, Alan Sheinbaum, Timothy C. Simmons, Rebecca Slomovic, Brennan M. Spiegel, Mitchell J. Spirt, James Sul and Rabindra R. Watson. Scheduled unsedated colonoscopy - a novel tool for managing no shows due to lack of escorts required for conscious sedation. Gastrointestinal Endoscopy, 2014-05-01, Volume 79, Issue 5, Pages AB178-AB179
- [Background] Terruzzi V, Meucci G, Radaelli F, Terreni N, Minoli G. Routine versus "on demand" sedation and analgesia for colonoscopy: a prospective randomized controlled trial. Gastrointest Endosc. 2001 Aug;54(2):169-74. doi: 10.1067/mge.2001.113923. PMID 11474385
- [Background] Leung FW, Harker JO, Jackson G, Okamoto KE, Behbahani OM, Jamgotchian NJ, Aharonian HS, Guth PH, Mann SK, Leung JW. A proof-of-principle, prospective, randomized, controlled trial demonstrating improved outcomes in scheduled unsedated colonoscopy by the water method. Gastrointest Endosc. 2010 Oct;72(4):693-700. doi: 10.1016/j.gie.2010.05.020. Epub 2010 Jul 8. PMID 20619405
- [Background] Leung JW, Mann SK, Siao-Salera R, Canete W, Leung FW. The established and time-tested water exchange method in scheduled unsedated colonoscopy significantly enhanced patient-centered outcomes without prolonging procedural times - A RCT. J Interv Gastroenterol. 2013;3(1):7-11.
- [Background] Hsieh YH, Koo M, Leung FW. A patient-blinded randomized, controlled trial comparing air insufflation, water immersion, and water exchange during minimally sedated colonoscopy. Am J Gastroenterol. 2014 Sep;109(9):1390-400. doi: 10.1038/ajg.2014.126. Epub 2014 Jun 3. PMID 24890443
- [Background] Cadoni S, Gallittu P, Sanna S, Fanari V, Porcedda ML, Erriu M, Leung FW. A two-center randomized controlled trial of water-aided colonoscopy versus air insufflation colonoscopy. Endoscopy. 2014 Mar;46(3):212-8. doi: 10.1055/s-0033-1353604. Epub 2013 Nov 11. PMID 24218307
- [Background] Cadoni S, Sanna S, Gallittu P, Argiolas M, Fanari V, Porcedda ML, Erriu M, Leung FW. A randomized, controlled trial comparing real-time insertion pain during colonoscopy confirmed water exchange to be superior to water immersion in enhancing patient comfort. Gastrointest Endosc. 2015 Mar;81(3):557-66. doi: 10.1016/j.gie.2014.07.029. Epub 2014 Sep 26. PMID 25262100
- [Background] Cadoni S, Falt P, Gallittu P, Liggi M, Mura D, Smajstrla V, Erriu M, Leung FW. Water Exchange Is the Least Painful Colonoscope Insertion Technique and Increases Completion of Unsedated Colonoscopy. Clin Gastroenterol Hepatol. 2015 Nov;13(11):1972-80.e1-3. doi: 10.1016/j.cgh.2015.04.178. Epub 2015 May 5. PMID 25956838
- [Background] Kim HG. Painless Colonoscopy: Available Techniques and Instruments. Clin Endosc. 2016 Sep;49(5):444-448. doi: 10.5946/ce.2016.132. Epub 2016 Sep 30. PMID 27744665
- [Background] Morgan J, Thomas K, Lee-Robichaud H, Nelson RL, Braungart S. Transparent cap colonoscopy versus standard colonoscopy to improve caecal intubation. Cochrane Database Syst Rev. 2012 Dec 12;12(12):CD008211. doi: 10.1002/14651858.CD008211.pub3. PMID 23235654
- [Background] Holme O, Bretthauer M, de Lange T, Seip B, Huppertz-Hauss G, Hoie O, Sandvei P, Ystrom CM, Hoff G. Risk stratification to predict pain during unsedated colonoscopy: results of a multicenter cohort study. Endoscopy. 2013 Sep;45(9):691-6. doi: 10.1055/s-0033-1344239. Epub 2013 Jul 24. PMID 23884794
- [Background] Wang L, Jia H, Luo H, Kang X, Zhang L, Wang X, Yao S, Tao Q, Pan Y, Guo X. A novel intubation discomfort score to predict painful unsedated colonoscopy. Medicine (Baltimore). 2021 Mar 12;100(10):e24907. doi: 10.1097/MD.0000000000024907. PMID 33725848
- [Background] Anderson JC, Gonzalez JD, Messina CR, Pollack BJ. Factors that predict incomplete colonoscopy: thinner is not always better. Am J Gastroenterol. 2000 Oct;95(10):2784-7. doi: 10.1111/j.1572-0241.2000.03186.x. PMID 11051348
- [Derived] Leung FW, Cheung R, Friedland S, Jacob N, Leung JW, Pan JY, Quan SY, Sul J, Yen AW, Jamgotchian N, Chen Y, Dixit V, Shaikh A, Elashoff D, Saha A, Wilhalme H. Prospective randomized controlled trial of water exchange plus cap versus water exchange colonoscopy in unsedated veterans. Gastrointest Endosc. 2025 Feb;101(2):402-413.e2. doi: 10.1016/j.gie.2024.07.010. Epub 2024 Jul 23. PMID 39053653

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects will be selected from patients scheduled for colonoscopy as part of their routine care. Eligible subjects will be asked to sign the ICF. Control and study methods will be explained, and study subjects will undergo a questionnaire, physical examination, and unsedated colonoscopy with the standard (control) or study methods. Ineligible patients will be offered unsedated colonoscopy by standard method, outside the research study.
Period: Overall Study
Arm/Group | Control Method | Study Method
Started | 137 | 143
Completed | 137 | 143
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All patients were US veterans scheduled for routine colonoscopy as part of their standard of care.
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Method | Study Method | Total
Number analyzed (Participants) | 137 | 143 | 280
Age, Categorical [Count of Participants; unit: Participants] — Male and female veterans aged 50-80, inclusive.
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 137 | 143 | 280
    >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 12
  Male | 132 | 136 | 268
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 18 | 34
  Not Hispanic or Latino | 120 | 124 | 244
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 7 | 7 | 14
  Native Hawaiian or Other Pacific Islander | 4 | 2 | 6
  Black or African American | 34 | 27 | 61
  White | 88 | 100 | 188
  More than one race | 2 | 5 | 7
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Count of Participants; unit: Participants] — All enrolled participants were United States Veterans
  Participants
    United States | 137 | 143 | 280

OUTCOME MEASURES:

1. Primary Outcome: Real Time Maximum Insertion Pain
Description: Pain during insertion reported to the unblinded assisting nurse, visual analogue scale, VAS: 0=none, 10=most severe. The highest pain score will be tabulated for analysis. Timing of data collection will be at the discretion of the nurse to minimize bias by colonoscopist behavior.
Time Frame: Insertion pain was measured during the duration of the colonoscopy procedure, which lasted on average for about 1 hour
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Method | Study Method
Number analyzed (Participants) | 137 | 143
score on a scale | 2.6 (2.4) | 2.9 (2.5)
Statistical Analysis 1: Comparison: Control Method vs Study Method; Chi Square; Test type: Superiority; p = 0.62, Chi-squared

2. Secondary Outcome: Proportion of Patients With No Insertion Pain
Description: Proportion of patients who report no pain during insertion of the colonoscope.
Time Frame: Pain was measured during the duration of the colonoscopy procedure, which lasted on average for about 1 hour
Measure: Count of Participants; unit: Participants
Arm/Group | Control Method | Study Method
Number analyzed (Participants) | 137 | 143
Participants | 38 | 41

3. Secondary Outcome: Insertion Time
Description: Time to cecum (clock display on monitor), faster insertion is a quality marker
Time Frame: Insertion time in minutes was measured during the duration of the colonoscopy procedure, which lasted on average for about 1 hour
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Control Method | Study Method
Number analyzed (Participants) | 137 | 143
Minutes | 18.8 (15.9) | 18.6 (15.6)

4. Secondary Outcome: Right Colon Adenoma Detection Rate (ADR)
Description: Right colon Adenoma Detection Rate (ADR) is the proportion of patients with at least one adenoma in the part of the colon between the cecum and the hepatic flexure.
Time Frame: Adenoma Detection Rate (ADR) was measured during the duration of the colonoscopy procedure, which lasted on average for about 1 hour
Measure: Count of Participants; unit: Participants
Arm/Group | Control Method | Study Method
Number analyzed (Participants) | 137 | 143
Participants | 40 | 27

ADVERSE EVENTS:
Time Frame: Adverse events and serious adverse event, were monitored for the total duration of the study, which was up to 30 days.
Description: Our definition of Adverse or Serious Adverse Events does not differ from the clinicaltrials.gov definitions.
  All colonoscopy procedures were routinely performed by gastroenterologists with at least 5 years of experience.
Arm/Group | Control Method | Study Method
All-Cause Mortality (participants affected / at risk) | 0/137 | 0/143
Serious Adverse Events (participants affected / at risk) | 0/137 | 0/143
Other Adverse Events (participants affected / at risk) | 0/137 | 0/143

LIMITATIONS AND CAVEATS:
The limitations included: (1) subjects were mostly male Veterans, (2) colonoscopists were unblinded, (3) colonoscopist-assessed patient anxiety was subjective and not measured on a standardized anxiety scale.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2017-08-14): https://cdn.clinicaltrials.gov/large-docs/59/NCT03160859/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-14): https://cdn.clinicaltrials.gov/large-docs/59/NCT03160859/SAP_001.pdf
  • Informed Consent Form (2019-12-16): https://cdn.clinicaltrials.gov/large-docs/59/NCT03160859/ICF_002.pdf